CLINICAL TRIAL: NCT06479057
Title: Integrating PROACTive Care Pathways to Empower and Support Cancer Patients (PROACT)
Brief Title: PROACT is a Prospective Master Protocol for a Cohort Study Focused on Evaluating the Implementation of Integrated Proactive Supportive Care Pathways at Gustave Roussy
Acronym: PROACT
Status: Recruiting | Type: Observational
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-A01225-40; 2023/3662 (Other: CSET number)
Record Dates: First submitted 2024-04-05; First posted 2024-06-27 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Any Cancer
Keywords: supportive care pathway; cancer; master protocol; supportive care; Distress
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PROACT Supportive Care pathways: This is a prospective cohort study including patients participating in institutional supportive care pathways at diagnosis, during treatment and after treatment.
  Interventions: Other: Supportive Care Pathway

INTERVENTIONS:
Other: Supportive Care Pathway — All pathways include a medical consultation with comprehensive needs assesment and evidence-based coordinated supportive care referrals at institutional and community-based level.

SUMMARY:
PROACT is a prospective master protocol for a cohort study focused on evaluating the implementation of integrated proactive pathways of supportive care.

This is an observational cohort study in the context of a quality-of-care initiative.

It will be evaluated by its impact on patient's distress measured by the NCCN's Distress thermometer at 12 weeks after entering the pathway.

DETAILED DESCRIPTION:
The primary study endpoint of PROACT is patient distress and supportive care needs (NCCN Distress Thermometer and NCCN Problem list) over a 12-week period after the supportive care needs assessment and referrals in the context of a PROACT pathway.

Secondary study endpoints include:

1. To evaluate the Reach of each pathway through the number of patients who participated in supportive care needs' assessment and in each supportive care intervention (administrative review of attendance log)
2. To evaluate the diversity of patients included in each pathways through evaluation of sociodemographic and economic profile (Socioeconomic and demographic self-reported questionnaire)
3. To evaluate the impact of each pathway and each supportive care intervention on patient's overall health status (EQ-E5-EL)
4. To evaluate the impact of each pathway and each supportive care intervention on patient's quality of life (EORTC QLQ C30)
5. To evaluate the impact of each pathway and each supportive care intervention on symptom burden (MDASI)
6. To evaluate the impact of each pathway and each supportive care intervention on anxiety (HADS)
7. To evaluate the impact of each pathway and each supportive care intervention on Insomnia levels (ISI)
8. To evaluate the impact of each pathway and each supportive care intervention on sexual health (EORTC SHQ-C22)
9. To evaluate the Physician's Adoption of each pathway through the proportion of physicians referring patients to the pathways (referral log)
10. To evaluate patient's adoption through the proportion of patients adhering to supportive care interventions as intended (attendance log)
11. To evaluate patient experience and satisfaction with the pathways (PACIC and adhoc satisfaction questionnaires.
12. To evaluate implementation in through a qualitative analyses of experience, implementation barriers and facilitators (focus groups with patients and providers)
13. To plan for Maintenance of the pathway through a cost effectiveness analysis.
14. To evaluate the impact of each pathway and each supportive care intervention on Intestinal Symptoms (LARS score). if indicated for the specific population
15. To evaluate the impact of each pathway and each supportive care intervention on Anal Incontinence (Wexner score). if indicated for the specific population
16. To evaluate the impact of each pathway and each supportive care intervention on Urinary Symptoms (USP score). if indicated for the specific population
17. To evaluate the impact of each pathway and each supportive care intervention on Hematologic Cancer (FACT-BMT)
18. To evaluate the impact of each pathway and each supportive care intervention on Montgomery Borgatta Caregiver Burden Scale. if indicated for the specific population.
19. To evaluate the healthcare professionals participating in the pathway to screen vulnerability and prevent treatment related burden (F-SUS)

This is a master protocol study that is conducted by collecting sub-studies for each supportive care intervention which share key design components and operational aspects leading to a higher level of coordination than the one achieved by independently conducted studies.

Methodology: it is a mix of quantitative and qualitative methods to assess the Reach, Efficacy and potential for Adoption, while identifying barriers to Implementation and strategies to Maintain the pathway in the institution guided by the RE-AIM framework. Data collection will allow evaluation in a macro level (integrated supportive care pathway including supportive care needs assessment and tailored multidisciplinary referrals) and in a micro level (separated for each supportive care intervention).

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of cancer (any cancer type, any stage)
* Age ≥ 18 years old
* Received an integrated supportive care need assessment.
* Sign the consent form for the PROACT study.

Exclusion Criteria:

* Absence or inability of written consent from the patient.
* Does not understand or speak French.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with any cancer type, any stage receiving supportive care interventions at Gustave Roussy.
  For the primary endpoint all the patients participating in supportive care pathways with formal supportive care needs assessment and targeted referrals will be invited to participate. For the secondary endpoints, any patient included in the supportive care interventions at the institution may participate.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2024-01-11 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Patient distress | over a 12-week period after the integrated supportive care needs assessment.
  Patient distress collected with NCCN Distress Thermometer
Patient unmet needs | over a 12-week period after the integrated supportive care needs assessment.
  Patient unmet needs collected with problem list from NCCN Distress thermometer

SECONDARY OUTCOMES:
Reach of the pathway | week 12
  Proportion of patients who accepted the supportive care needs assessment (descriptive numbers from attendance log)
Diversity of pathway participants | week 12
  Socioeconomic characteristics of participants in the pathway measure by a self-reported socioeconomic questionnaire
Impact of the pathway in overall health status | week 12, and 24
  Overall health status measured by the EQ-ED-5L
Impact of the pathway in Quality of life | week 12, and 24
  Quality of life measured by the EORTC QLQ C30
Impact of the pathway in symptom burden | week 12, and 24
  Symptom burden measured by the MDASI Questionnaire.
Impact of the pathway on anxiety levels | week 12, and 24
  Anxiety measured by HADS
  * only for patients reporting anxiety at baseline
Impact of the pathway on insomnia levels | week 12, and 24
  Insomnia measured by ISI
  *only for patients reporting insomnia at baseline
Impact of the pathway on sexual health | week 12, and 24
  Sexual health measured by EORTC SHQ-C22
  *only for patients reporting sexual dysfunction at baseline
Adoption of Physician | week 12
  Proportion of physicians referring patients to the supportive care pathway (descriptive numbers from referral logs)
Adoption of Patient | week 12
  Proportion and of patients that fully adopted each supportive care intervention (e.g.; in the after cancer pathway: attendance to consultations/seminaries/classes, completion of a supportive care program, usage data for Resilience app).
Patient Experience | week 12
  Patient experience measured by the PACIC questionnaire.
Patient Satisfaction with the pathway | week 12
  Patient satisfaction measured by an ad hoc satisfaction questionnaire
Provider Experience - Qualitative evaluation | week 12
  Focus groups with healthcare providers to explore overall experience, workload and implementation challenges
Patient Satisfaction/Experience - Qualitative evaluation | week 12
  Focus groups with patient to explore overall experience and implementation challenges
Maintenance of the pathway through a cost effectiveness analysis (QALYs) | week 12
  Maintenance of the pathway through a cost effectiveness analysis. Costs from the perspective of the French national health insurance will be assessed during the study period. This will be calculated by administrative data review of internal allocated resources for pathway delivery and estimated costs of use of hospital services (unplanned hospitalization, consultations, and emergency visits recorded in the electronic medical records).
  QALYs (quality-adjusted life years) will be measured using utility values derived from the EuroQol-5D (EQ-5D-5L) (https://euroqol.org/) for French general population (Andrade et al. PharmacoEconomics 2020). QALYs will be computed combining survival time by utility values.
Impact of the pathway on Intestinal Symptom | week 24
  Intestinal Symptoms measured by LARS score.
  *only for patients with digestive cancer
Impact of the pathway on Anal incontinence | week 24
  Anal incontinence measured by Wexner score.
  *only for patients with digestive cancer
Impact of the pathway on Urinary symptoms | week 24
  Urinary symptoms measured by USP score.
  *only for patients with digestive cancer
Impact of the pathway on Functional Assessment of Cancer Therapy-Bone Marrow Transplant | week 12, week 24
  Functional Assessment of Cancer Therapy-Bone Marrow Transplant measured by FACT-BMT score.
  *only for patients with Hematologic Cancer
Impact of the pathway on caregiver burden | week 12
  Caregiver burden measured by Montgomery Borgatta Caregiver Burden Scale.
Impact of the pathway on healthcare professionals participating in the pathway to screen vulnerability and prevent treatment | week 12
  Healthcare professionals measured by F-SUS Score

CONTACTS AND LOCATIONS:
Overall Officials: Ines VAZ LUIS, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Gustave Roussy, Villejuif, France

REFERENCES:
- [Derived] Franzoi MA, Santolaya C, Martin E, Fasse L, Rouby P, Minot-This MS, Di Meglio A, Vaz-Luis I. "Let's talk about risk": co-designing a pathway to assess, communicate and act on individual risk of long-term toxicities after breast cancer. J Cancer Surviv. 2025 Jun 12. doi: 10.1007/s11764-025-01826-0. Online ahead of print. PMID 40504480
- [Derived] Franzoi MA, Pages A, Papageorgiou L, Di Meglio A, Laparra A, Martin E, Barbier A, Renvoise N, Arvis J, Scotte F, Vaz-Luis I. Evaluating the Implementation of Integrated Proactive Supportive Care Pathways in Oncology: Master Protocol for a Cohort Study. JMIR Res Protoc. 2024 Aug 26;13:e52841. doi: 10.2196/52841. PMID 39186774